CLINICAL TRIAL: NCT03197363
Title: Bialystok PLUS - Polish Longitudinal University Study
Brief Title: Białystok PLUS - Polish Longitudinal University Study
Acronym: Bialystok+
Status: Enrolling by invitation | Type: Observational
Sponsor: Medical University of Bialystok (Other)
Collaborators: University Medicine Greifswald (Other); City of Białystok (Unknown); Marshall's Office of Podlaskie Voivodship (Unknown)
Responsible Party: Sponsor
Other Study IDs: B+
Record Dates: First submitted 2017-06-20; First posted 2017-06-23 (Actual); Last update posted 2023-03-15 (Actual); Status verified 2023-03

CONDITIONS: Cardiovascular Diseases; Diabetes; Neuro-Degenerative Disease; Obesity; Pulmonary Disease; Neoplastic Disease
Keywords: Civilization diseases; Cardiovascular Risk Factor; Population study; Intestinal microbiome; Oral microbiome
MeSH Terms: conditions — Cardiovascular Diseases; Diabetes Mellitus; Obesity; Lung Diseases; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples: Serum, plasma (will be collected from fasting blood samples) In this study we will be isolated Peripheral Blood Mononuclear Cells (PBMC) from fresh blood sampled on EDTA as anticoagulant.
  Saliva samples (unstimulated and stimulated) Urine samples Stool samples (for analysis intestinal microbiome)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Białystok PLUS: Participation in the study will be offered to 10000 inhabitants of Bialystok aged 20-80 years. They will be randomly selected from the registry of Bialystok inhabitants. The goal of study is to discover novel risk factors and mechanisms underlying civilization diseases.
  Interventions: Other: Discovering novel risk factors.

INTERVENTIONS:
Other: Discovering novel risk factors. — The study protocol includes multiple imaging and functional investigations (including heart, carotid, thyroid, liver ultrasound, fundoscopy, plethysmography, pulse wave velocity, ankle-brachial index, ECG, body composition measured by bioimpedance and dual energy x-ray absorptiometry, anthropometric assessment, rhinometry, hand grip test, oral glucose tolerance test, advance glycation end-products measurement, voice recording. There will be a detailed and verified questionnaires concerning various activities of the subject: physical activity, depression, sino-nasal symptoms, prostate hypertrophy, female urinary tract symptoms, quality of life, smoking and drinking addiction, hirsutism.

SUMMARY:
The main goal of the study is to provide a unique multidimensional picture of the health of the population with simultaneous optimal standards of sampling, processing and storing of data and biomaterial that will allow discovering novel mechanisms in the development and progression of common civilization diseases. In the effect it will improve prevention, diagnosis and treatment.

DETAILED DESCRIPTION:
One of the objectives of this project is to obtain comprehensive information on the health status (including subclinical disorders), genomics, risk factors, health behavior and sociodemographic data from large, representative sample of population of Białystok city inhabitants.

The study will assess many systems, the major emphasis will be given to the most common diseases associated with modern lifestyle (civilization diseases): cardiovascular, metabolic and endocrine, neurodegenerative, neoplastic and pulmonary. There are many interactions between them that might be missed when not analyzed together. Apart from those most common diseases we will also asses others, including allergies, airway dysfunction - both upper and lower, urinary incontinency, gastrointestinal disorders, eye diseases. There may be many common underlying mechanisms of the diseases that now seem to be distant and independent, because of insufficient knowledge.

Health status assessment will refer to many areas of medicine and will include clinical data, medical images, as well as biological samples and voice recording samples. We plan to combine imaging (fundoscopy, ultrasound examinations of heart, vessels, thyroid, liver) with state of the art functional studies (AGE measurement, pulse wave velocity, central pressure, plethysmography with the analysis of diffusing capacity of lung for carbon monoxide and NO concentration, spiroergometry, oral glucose tolerance test.

Voice samples will be analyzed in the speech analysis software, it will help in the diagnosis of civilization diseases such as diabetes, depression, and atherosclerosis.

Participants will fill in detailed questionnaires that will provide information about their family history, dietary habits, socioeconomic status, stress coping strategies, lifestyle, exposure to harmful environment, various symptoms, history of diagnosed diseases and treatment.

The study is designed as prospective, so in the future, additional information on occurrence of diseases or deaths will allow to estimate disease incidence, morbidity or mortality in studied population.

ELIGIBILITY:
Inclusion Criteria:

* inhabitants of Bialystok (randomly selected from the registry of Bialystok inhabitants)
* age 20-80

Exclusion Criteria:

* disagreement of the invited person

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Inhabitants of Bialystok (selected from the registry of Bialystok inhabitants). Stratified sampling will be performed, based on sex and age strata (10-year intervals) in order the sample to be representative for gender and age distribution in Bialystok population.
Sampling Method: Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2018-11-05 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Death or the occurrence of diseases | 5 years
  Death or the occurrence of diseases: cardiovascular diseases, diabetes, neuro-degenerative diseases, obesity, pulmonary diseases, neoplastic diseases

CONTACTS AND LOCATIONS:
Overall Officials: Karol A. Kaminski, Professor, Principal Investigator — Medical University of Bialystok
Locations (1):
- Medical University of Bialystok, Bialystok, Poland

IPD SHARING:
Plan to Share IPD: Yes
Scientists and researchers who collaborate on Bialystok PLUS study organization have access to results of examinations and analyses of biological material. Personal data are protected and only designated persons have access to them.

REFERENCES:
- See also: This page contains information about Bialystok PLUS study. — http://bialystok.plus/